CLINICAL TRIAL: NCT02627794
Title: Rates of Middle Meatus (MM) Synechiae Formation Post Endoscopic Sinus Surgery (ESS): A Double-blind Randomized Controlled Study Comparing Silastic and Restora™ Steroid Eluting MM Spacer
Brief Title: Rates of Middle Meatus Synechiae Formation Post Endoscopic Sinus Surgery
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to financial issues of Restora spacer company.
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Martin L. Hopp, MD, Principal Investigator, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00039737
Record Dates: First submitted 2015-12-07; First posted 2015-12-11 (Estimated); Results first posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-10

CONDITIONS: Sinusitis
Keywords: Middle Meatus; Synechiae; Endoscopic Sinus Surgery; Silastic spacer; Restora™ steroid eluting MM spacer
MeSH Terms: conditions — Sinusitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Silastic Silicone & Restora™ Steroid eluting spacer (Experimental): Silastic Silicone spacers are actively being used as the standard of care.
  Restora™ Steroid eluting spacer (experimental).
  Each nostril will receive one each of above spacers.
  Interventions: Device: Restora™ Steroid eluting spacer; Device: Silastic Silicone Spacer

INTERVENTIONS:
Device: Restora™ Steroid eluting spacer — The Restora™ Steroid eluting spacer will be inserted into the middle meatal space after surgery. The spacer will be left in the middle meatus for a period of 6-8 days following surgery.
  Other Names: Experimental arm
Device: Silastic Silicone Spacer — The Silastic Silicone Spacer will be inserted into the middle meatal space after surgery. The spacer will be left in the middle meatus for a period of 6-8 days following surgery.
  Other Names: Control Arm

SUMMARY:
Endoscopic sinus surgery (ESS) is the gold standard surgical intervention for chronic rhinosinusitis that is not adequately controlled with maximal medical therapy.

In some patients, underlying inflammation (discharge, edema and polyposis), compounded by inflammation caused by surgical trauma may lead to an uncontrolled healing response, which results in the synechiae formation in the middle meatus (MM).

Incidence of synechiae formation varies in literature and ranges between 4-35%. Presence of middle meatal synechiae can impair sinus drainage, promote sinusitis, and limit endoscopic visualization of the sinus cavities postoperatively. This may result in difficulty in performing postoperative routine endoscopic debridement and examination, which is paramount to a successful outcome from ESS. Spacers are often inserted during surgery between nasal mucosal surfaces to prevent synechiae.

The aim of this study is to see if a steroid-impregnated spacer is more effective at reducing inflammation after sinus surgery than a Silastic spacer.

DETAILED DESCRIPTION:
Endoscopic sinus surgery (ESS) is the gold standard surgical intervention for chronic rhinosinusitis that is not adequately controlled with medical therapy. Synechiae formation in the middle meatus is the most common complication of endoscopic sinus surgery. Synechiae describes the adhesion of two opposing mucosal surfaces in the nasal cavity that can cause scarring and obstruction of the nasal passage. Incidence of synechiae formation varies in literature and ranges between 4-35 %. Presence of middle meatal synechiae can impair sinus drainage, promote sinusitis, and limit endoscopic visualization of the sinus cavities postoperatively. This may result in difficulty in performing postoperative routine endoscopic debridement and examination, which is paramount to a successful outcome from ESS.

To prevent synechiae formation, numerous studies have been published evaluating the effectiveness of absorbable and non-absorbable spacers placed in the middle meatus for 1-2 weeks postoperatively. The spacer is meant to prevent contact between the denuded surfaces of the middle turbinate and the lateral nasal wall during re-epithelialization. In general, non-resorbable spacers that have been used include sponges, cotton gauze and plastic sheets. Of these, Silastic Silicone sheets have been used in a number of hospitals across the US and Canada. Lee and Baguley have demonstrated the effectiveness of Silastic spacers in reducing the risk of synechiae formation to between 0-6 %. There are also a number of resorbable spacers that are in use, which are preferred by some physicians because there is minimal need to remove the packing materials as they naturally are removed or resorbed during the healing period.

In a recent meta-analysis, Lee et al has revealed that usage of middle meatal spacers (absorbable and non-absorbable) did not decrease the rate of synechiae formation to a statistically significant degree compared to not using any spacer. However, when subgroup analysis was performed, non-absorbable spacer usage demonstrated a statistically significant lower incidence of synechiae compared to no spacers. This can be explained in part by an inherent capability of the absorbable spacer material to degrade to smaller size particulates that, if caught in the healing tissue, could illicit local inflammatory response to slow down the healing and cause further synechiae formation. This mechanism was demonstrated by Maccabee et al in a rabbit model, where fibers of the absorbable spacer became incorporated into healing mucosa and increased the extent of the inflammatory response and formation of fibrosis.

To improve outcomes, physicians have attempted to load steroids such as Triamcinolone and antibiotics such as Neosporin into nasal packing and/or stents. However, residence of the drug in the intended treatment space is minimized as the drug, which is not bound to the spacer, quickly releases and may not remain long enough to impact inflammatory response. A Mometasone Furoate coated stent (Propel™), manufactured by Intersect ENT, is currently the only drug coated nasal stent that has a claim of longer sustained release. In a randomized, controlled, double-blind trial, Marple et al found that this Mometasone Furoate steroid-eluting bio-absorbable stent could significantly improve postoperative outcomes compared to a non-steroid eluting placebo arm with the same stent. Zhao et al conducted a systematic review of the efficacy of this steroid-eluting stent (Propel) vs inert (both resorbable and non-resorbable) spacers and again confirmed that there are lower rates of synechiae formation in the steroid-eluting treatment groups. However, anecdotal evidence, based on discussion with a number of surgeons in the field, suggests that a drug-loaded resorbable spacer may be subject to the same issues as non-drug-loaded resorbable spacers, namely late stage degradation of the material that can cause a secondary spike of the inflammatory cascade, requiring additional surgical intervention to remove the remaining debris.

Therefore, it has been hypothesized that a steroid eluting non-absorbable spacer may provide optimal benefit for the patient's outcome. The Restora™ spacer is made of a biocompatible non-resorbable material that is expected to deliver up to 370 µg of Mometasone Furoate. The steroid elutes out of the spacer and onto the surrounding mucosal tissue during the 6-8 day period during which it is retained.

This study is designed to evaluate basic device usability and confirm safety and effectiveness of the Restora™ Steroid eluting spacer as compared to the standard of care Silastic Silicone spacer.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years
2. Diagnosis of chronic rhinosinusitis (CRS), per current guidelines
3. Patients who need to undergo primary bilateral complete endoscopic sinus surgery
4. Subject has the ability to follow the study instructions, is willing to be available on the specific required study visit days, and is willing to complete all study visit procedures and assessments
5. Subject must understand the research nature of this study and sign an informed consent prior to the performance of any study-specific procedure or assessment

Exclusion Criteria:

1. Subject is pregnant or breast feeding
2. Patients with sino-nasal tumors
3. Patients solely undergoing nasal septal reconstruction
4. Patients with previous history of endoscopic sinus surgery
5. Cystic fibrosis or syndromic patients
6. Patients with autoimmune diseases
7. Patients who have taken oral steroids less than 30 days prior to surgery
8. Patients with a history or diagnosis of glaucoma or ocular hypertension
9. Any other circumstance or condition that in the Investigator's opinion causes the subject to be an inappropriate candidate for participating in this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin L Hopp, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: nasal
Groups:
- Restora™ Steroid Eluting & Silastic Silicone Spacers: This study arm receives both the experimental treatment, a Restora™ Steroid eluting spacer and Silastic Silicone spacer.
  Both spacers will be inserted into the middle meatal space after surgery. The spacer will be left in the middle meatus for a period of 6-8 days following surgery.
Period: Overall Study
Arm/Group | Restora™ Steroid Eluting & Silastic Silicone Spacers
Started | 3; 6 nasal
Completed | 3; 6 nasal
Not Completed | 0; 0 nasal

BASELINE CHARACTERISTICS:
Population: Each participant received a Restora Spacer on one nostril and a silicone spacer on the other nostril. We had 3 participants in total, but each received two spacers.
Units Other Than Participants: Nose
Groups:
- Restora™ Steroid Eluting & Silastic Silicone Spacer: This arm receives both Restora™ Steroid eluting & Silastic Silicone spacers.
  The Restora™ Steroid eluting and Silastic Silicone Spacers will be inserted into the middle meatal space after surgery. The spacer will be left in the middle meatus for a period of 6-8 days following surgery.
Arm/Group | Restora™ Steroid Eluting & Silastic Silicone Spacer
Number analyzed (Participants) | 3
Number analyzed (Nose) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Middle Meatal Synechiae After Endoscopic Sinus Surgery in Silastic and Restora Steroid Eluting Spacer.
Description: The main objective of the trial is to evaluate basic device usability and confirm safety and effectiveness of Restora™ Mometasone Furoate eluting spacer as compared to a Silastic spacer. 35-day sinonasal mucosal inflammation will be assessed by rigid endoscopy and graded on Lund-Kennedy sinus mucosal endoscopic staging system.
Time Frame: Participants will be followed for the duration of post op standard of care, an expected average of 90 days.
Measure: Count of Participants; unit: Participants
Groups:
- Silastic Silicone Spacer: Silastic Silicone spacers are actively being used as the standard of care.
  Silastic Silicone Spacer: The Silastic Silicone Spacer will be inserted into the middle meatal space after surgery. The spacer will be left in the middle meatus for a period of 6-8 days following surgery.
- Restora™ Steroid Eluting Spacer: This study arm receives the experimental treatment, a Restora™ Steroid eluting spacer.
  Restora™ Steroid eluting spacer: The Restora™ Steroid eluting spacer will be inserted into the middle meatal space after surgery. The spacer will be left in the middle meatus for a period of 6-8 days following surgery.
Arm/Group | Silastic Silicone Spacer | Restora™ Steroid Eluting Spacer
Number analyzed (Participants) | 3 | 3
Participants | 3 | 3

2. Secondary Outcome: 90-day Sinonasal Mucosal Inflammation Assessment
Description: 90-day sinonasal mucosal inflammation assessed by rigid endoscopy and graded on Lund-Kennedy sinus mucosal endoscopic staging system
Time Frame: Participants will be followed for the duration of post op standard of care, an expected average of 90 days.
Population: Zero participants were analyzed as data were not significant (not enough data); Study closed prior to being able to enroll sample size (N=50) goal.
Arm/Group | Restora™ Steroid Eluting & Silastic Silicone Spacer
Number analyzed (Participants) | 0

3. Secondary Outcome: 35 and 90-day Intraocular Pressure (IOP) Assessment
Description: 35 and 90-day intraocular pressure (IOP) assessed using applanation tonometry and compared to baseline IOP obtained preoperatively
Time Frame: Participants will be followed for the duration of post op standard of care, an expected average of 90 days.
Population: as for outcome 2
Arm/Group | Restora™ Steroid Eluting & Silastic Silicone Spacer
Number analyzed (Participants) | 0

4. Secondary Outcome: 35 and 90-day Post ESS Incidence of Middle Meatal Synechiae
Description: 35 and 90-day post ESS incidence of middle meatal synechiae
Time Frame: Participants will be followed for the duration of post op standard of care, an expected average of 90 days.
Population: as for outcome 2
Arm/Group | Restora™ Steroid Eluting & Silastic Silicone Spacer
Number analyzed (Participants) | 0

5. Secondary Outcome: 90-day Sinonasal Outcomes Test-22 (SNOT- 22) Scores
Description: 90-day Sinonasal Outcomes Test-22 (SNOT- 22) scores
Time Frame: Participants will be followed for the duration of post op standard of care, an expected average of 90 days.
Population: as for outcome 2
Arm/Group | Restora™ Steroid Eluting & Silastic Silicone Spacer
Number analyzed (Participants) | 0

6. Secondary Outcome: 35-day Frequency of Postoperative Interventions
Description: 35-day frequency of postoperative interventions, including lyses of adhesions and debridement.
Time Frame: Participants will be followed for the duration of post op standard of care, an expected average of 90 days.
Population: as for outcome 2
Arm/Group | Restora™ Steroid Eluting & Silastic Silicone Spacer
Number analyzed (Participants) | 0

7. Secondary Outcome: 35-day Frequency of Oral Steroid Rescue
Description: 35-day frequency of oral steroid rescue
Time Frame: Participants will be followed for the duration of post op standard of care, an expected average of 90 days.
Population: as for outcome 2
Arm/Group | Restora™ Steroid Eluting & Silastic Silicone Spacer
Number analyzed (Participants) | 0

8. Secondary Outcome: 35 Days Middle Turbinate Position
Description: 35 days middle turbinate position
Time Frame: Participants will be followed for the duration of post op standard of care, an expected average of 90 days.
Population: as for outcome 2
Arm/Group | Restora™ Steroid Eluting & Silastic Silicone Spacer
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Silastic Silicone Spacer | Restora™ Steroid Eluting Spacer
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-18): https://cdn.clinicaltrials.gov/large-docs/94/NCT02627794/Prot_SAP_000.pdf